CLINICAL TRIAL: NCT01519609
Title: Double Blind Randomised Trial Comparing Moviprep and Phosphoral as Bowel Prep Before
Brief Title: Trial Comparing Moviprep and Phosphoral as Bowel Prep Before Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Thorbjorn Sommer, M.D, Ph.D Associate Professor, Randers Regional Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Randers-Moviprep
Record Dates: First submitted 2011-09-16; First posted 2012-01-27 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Cancer
Keywords: Bowel prep; Safety; Efficacy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moviprep (Active Comparator): Moviprep bowel preb
  Interventions: Drug: bowel prep before endoscopy
- Phosphoral (Active Comparator): Bowel prep
  Interventions: Drug: bowel prep before endoscopy

INTERVENTIONS:
Drug: bowel prep before endoscopy — bowel prep before colonoscopy

SUMMARY:
Using Moviprep patients use shorter time to do a bowel prep before colonoscopy. No major single center has docuemted the advantage of using moviprep as bowel prep before colonoscopy.This randomised study was conducted to compare moviprep with the present standard: Phosphoral to investigate the degree of bowel cleasing before colonoscopy in patients suspected of colorectal cancer, and to investigate number of days where patients need to stay home.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of colorectal cancer scheduled for colonoscopy

Exclusion Criteria:

* Patients with previous colorectal surgery
* Colonis Stenosis
* ASA > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Degree of bowel cleansing | 1 Day of colonoscopy
  Will be estimated by the patients and the colonoscopist

CONTACTS AND LOCATIONS:
Overall Officials: thorbjorn sommer, ph.D, Study Director — unaffilated
Locations (1):
- Randers Regions Hospital, Randers, Denmark